CLINICAL TRIAL: NCT03610152
Title: Does a Theory-Based Intervention to Improve Accountability Reduce Low-Value Preoperative Investigations in Patients Undergoing Ambulatory Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-5108
Record Dates: First submitted 2018-05-23; First posted 2018-08-01 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Low-value Pre-operative Investigations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Hospitals made aware of Choosing Wisely Canada recommendations and Health Quality Ontario data.
- Hospital wide policy (Experimental): A hospital-wide policy will be implemented whereby medically necessary preoperative tests for patients undergoing ambulatory surgery will be ordered at the discretion of the consulting anesthesiologists based on their clinical assessment of the patient.
  Interventions: Behavioral: Hospital Policy change

INTERVENTIONS:
Behavioral: Hospital Policy change — Implementation of a hospital wide policy whereby medically necessary preoperative tests for patients undergoing ambulatory surgery will be ordered at the discretion of the consulting anesthesiologist based on their clinical assessment of the patient.
  Arms: Hospital wide policy

SUMMARY:
The Institute of Medicine (IOM) suggests that up to 30% of healthcare is considered low-value, defined as 'a test or treatment for which there is no evidence of benefit to the patient or where there is evidence of more harm than benefit'. The investigators have previously found that more than 31% of Ontario patients, who go home the same day as their surgery, receive unnecessary cardiac testing and/or chest x-rays. In addition, the investigators identified an almost 30-fold variability in how tests are ordered between different hospitals. While identification of low-value care is an important first step, additional efforts are required to reduce this waste. The investigators previously explored the reasons behind low value test ordering through a qualitative study of surgeons and anesthesiologists. This work has informed the development of a theory-based intervention to reduce wasteful ordering. The proposed project will conduct a hospital level randomized controlled trial to determine if preoperative testing ordered by anesthesiologist and supported by a focused implementation strategy can decrease the use of low-value investigations before elective surgery where patients will go home the same day.

DETAILED DESCRIPTION:
The Institute of Medicine's (IOM) quality improvement framework includes the three pillars of underuse, overuse and misuse, though misuse and underuse have largely been the historical focus of quality improvement efforts (1). More recently, there is increasing recognition of the problem of overuse relating to "low-value care", defined as 'a test or treatment for which there is no evidence of patient benefit or where there is evidence of more harm than benefit'. The IOM suggests that as much as 30% of healthcare qualifies as low-value, which can lead to: poor patient outcomes due to adverse events of treatments or secondary unwarranted tests (with potential for over-treatment of incidental findings); and inefficient use of scarce healthcare resources threatening the sustainability of healthcare systems. In the context of Ontario, this would equate to over $15 billion wasted on low-value care in 2014 representing a major threat to the sustainability of the Ontario healthcare system. Unfortunately, recent studies have demonstrated similar levels of low-value care in Ontario currently, and suggest that there are considerable opportunities to reduce this waste within the province. For example, the investigators found previously that approximately 30% of patients received unnecessary cardiac testing and/or chest x-rays prior to ambulatory surgery (with almost 30-fold variability in ordering between institutions) (2,3).

Within Canada, provincial governments have made reducing low-value care a priority. Choosing Wisely Canada (CWC) (4,5) is a professionally led campaign to rally the medical professional to address this issue and make declarative statements about low-value care that physicians and patients should avoid or question across a broad range of specialties. To date, 37 Canadian medical specialty societies have developed over 150 recommendations pertaining to unnecessary tests, treatments and procedures.

Whilst the identification of potential areas of low-value care is an important first step in addressing this problem, additional efforts are required to ensure implementation of CWC recommendations. Before now, internationally and in Canada, the issue of implementing Choosing Wisely like recommendations has not received adequate attention. This project directly addresses this key priority for healthcare systems bringing together Ontarian experts from CWC, implementation science, relevant clinical content areas and knowledge users to develop and evaluate programs to implement CWC recommendations. The investigators will use state-of-the-art approaches from implementation science to develop and evaluate a major initiative to reduce low-value care in Ontario. Knowledge users include Health Quality Ontario, the Ontario Hospital Association and Choosing Wisely Canada.

ELIGIBILITY:
Inclusion Criteria:

• Hospitals in the 26th - 100th percentile for routine preoperative tests

Exclusion Criteria:

• Hospitals in the 0 - 25th percentile for routine preoperative tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Low-value preoperative investigations received | 12-months
  The proportion of patients that receive low-value preoperative investigations such as ECG, EKG, Chest X-Rays and chest stress testing within 60-days before surgery at each enrolled institution. Pooled data will be collected from administrative data source.

SECONDARY OUTCOMES:
Overnight admissions | 12-months
  Hospital rates of overnight admissions
Re-operation in 24-hours | 12-months
  Hospital rates of re-operation in 24 hours
All-cause mortality from the date of surgery | 12-months
  Hospital rates of 30-day all-cause mortality from the date of surgery
Patients who receive ECG, EKG, Chest X-ray and Cardiac stress test | 12-months
  The proportion of patients receiving each of the above pre-operative tests individually

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kirkham, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No